CLINICAL TRIAL: NCT03059537
Title: Validation of Stimulated ∆FGF19 for Diagnosing Bile Acid Diarrhoea
Acronym: VABAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lars Kristian Munck (Other)
Responsible Party: Sponsor-Investigator, Lars Kristian Munck, DMSci, Zealand University Hospital
Organization: Zealand University Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SJ-546
Record Dates: First submitted 2017-02-02; First posted 2017-02-23 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Bile Acid Malabsorption

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stimulation Test (Experimental): Study meal plus chenodeoxycholic acid: 1,250 mg single dose stimulation
  Interventions: Drug: Oral chenodeoxycholic acid stimulation

INTERVENTIONS:
Drug: Oral chenodeoxycholic acid stimulation — oral intake of chenodeoxycholic acid to stimulate the ileal bile acid transporter and farnesoid X receptor
  Other Names: Chenodeoxycolic acid

SUMMARY:
This study aims to validate a possible diagnostic test for bile acid diarrhoea prospectively compared to the SeHCAT scintigraphy. Fasting participants are given a standard meal and 1,250 mg chenodeoxycholic acid. The investigators measure fasting FGF19, bile acids species including 7-alpha-CHO and serial blood samples after the stimulation.

ELIGIBILITY:
Inclusion Criteria:

- Consecutive patients referred for SeHCAT

Exclusion Criteria:

* Treatment with sequestrants within one week before the SeHCAT.
* Treatment with any constipants/laxatives one day before the SeHCAT, with the exception of opioids, if the dosis has been stable in the prior 2 weeks.
* Pregnancy, screening by pregnancy test before inclusion.
* Breastfeeding women.
* Small bowel resection, including right sided hemicolectomy.
* Any ongoing treatment for inflammatory bowel disease with systemic steroids (i.e. budesonide or prednisone) or treatment in the prior 4 weeks.
* Allergies to constituents of Xenbilox: (chenodeoxycholic acid, cornflour, magnesium stearate, highly dispersed silica, gelatine, sodium dodecylsulphate, titanium dioxide (E171), quinolone yellow (E104), erythrosine (E127)
* Chronic or acute cholecystitis.
* Liver cirrhosis,
* Obstructed bile flow causing jaundice or elevated p-bilirubin (> 1,5 UNL).
* Known disability in gall bladder contractility.
* Bile duct atresia.
* Frequent gallstone attacks (>2/month).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-03-13 (Actual); Primary Completion 2017-11-27 (Actual); Study Completion 2017-11-27 (Actual)

PRIMARY OUTCOMES:
Negative predictive value of stimulated deltaFGF19 | Individual data are collected within one week
  For screening purposes for bile acid diarrhoea. Negative Predictive Value by Receiver Operating Curve analysis for SeHCAT < 10 %

SECONDARY OUTCOMES:
Other diagnostic and Nosographic propabilities stimulated deltaFGF19, SeHCAT < 10% | Individual data are collected within one week
  Positive predictive value, sensitivity and specificity for bile acid diarrhoea judged by FGF19 for SeHCAT <10%
Other diagnostic and Nosographic propabilities stimulated deltaFGF19, SeHCAT < 5% | Individual data are collected within one week
  Positive predictive value, sensitivity and specificity for bile acid diarrhoea judged by FGF19 for SeHCAT <5%
Diagnostic and Nosographic propabilities of 7alpha-CHO for SeHCAT <10% | Individual data are collected within one week
  Positive predictive value, sensitivity and specificity for bile acid diarrhoea judged by 7alpha-CHO for SeHCAT <10%
Diagnostic and Nosographic propabilities of 7alpha-CHO for SeHCAT <5% | Individual data are collected within one week
  Positive predictive value, sensitivity and specificity for bile acid diarrhoea judged by 7alpha-CHO for SeHCAT <5%
Correlation of FGF19 to clinical diarrhoea | Individual data are collected within one week
  Correlation of FGF19 (fasting and stimulated deltaFGF19) to diarrhoea by stool diary
Correlation of 7alpha-CHO to clinical diarrhoea | Individual data are collected within one week
  Correlation of fasting 7alpha-CHO to diarrhoea by stool diary
FGF19 by SeHCAT stratum | Individual data are collected within one week
  Median stimulated ∆FGF19 in SeHCAT stratum: 0-5%, >5.1-10%, >10.1-15%, > 15.1%.
7alpha-CHO by SeHCAT stratum | Individual data are collected within one week
  Median fasting 7alpha-CHO in SeHCAT stratum: 0-5%, >5.1-10%, >10.1-15%, > 15.1%.

CONTACTS AND LOCATIONS:
Overall Officials: Christian Borup, MD, Principal Investigator — Zealand University Hospital
Locations (5):
- Denmark (5):
  - Aalborg University Hospital, Aalborg
  - Aarhus University Hospital, Aarhus
  - Zealand University Hopsital, Holbæk
  - Hvidovre University Hospital, Hvidovre
  - Zealand University Hospital, Køge

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Borup C, Wildt S, Rumessen J, Graff J, Bouchelouche PN, Andersen TB, Vinter-Jensen L, Zaremba A, German Jorgensen SP, Gregersen T, Nojgaard C, Timm HB, Rainteau D, Gauliard E, Munck LK. Biochemical Diagnosis of Bile Acid Diarrhea: Prospective Comparison With the 75Seleno-Taurohomocholic Acid Test. Am J Gastroenterol. 2020 Dec;115(12):2086-2094. doi: 10.14309/ajg.0000000000000772. PMID 32740083